CLINICAL TRIAL: NCT01769560
Title: MeFirst: A Tailored Intervention to HPV Vaccine Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Vanessa K. Dalton, Associate Professor, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00069032
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Human Papillomavirus-Related Carcinoma
Keywords: tailored intervention; college aged students; HPV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Centers for Disease Control and Prevention (CDC) Fact Sheet (No Intervention): Participants will receive the CDC Fact sheet about HPV vaccination while they are taking the survey.
- MeFirst Intervention (Experimental): Participants will receive a tailored website regarding their own individualized risk for HPV and information about HPV Vaccination while they are taking the survey as opposed to receiving the CDC fact sheet. This tailored website is generated based on answers provided by each subject in the baseline survey.
  Interventions: Behavioral: MeFirst Tailored Intervention

INTERVENTIONS:
Behavioral: MeFirst Tailored Intervention — Participants will be lead through MeFirst, an interactive web-based tool that is tailored to their responses during the survey. This tool provides information regarding HPV Vaccination.
  Arms: MeFirst Intervention

SUMMARY:
This study will test whether a tailored, online educational intervention increases HPV vaccine uptake and intent among female college students.

DETAILED DESCRIPTION:
MeFirst is the first web-based, online, educational tool designed to promote Human Papillomavirus (HPV) vaccine awareness and understanding in an effort to improve HPV vaccine intent and uptake among female university students. HPV is the most common sexually transmitted infection and causes genital warts and cancer. The HPV vaccine has been recommended for girls ages 11-26 since 2006, yet vaccination rates remain low. Tailored online interventions may be more effective tools to promote behavior change among college students than traditional static interventions. The proposed study is a randomized controlled trial testing the efficacy of the MeFirst tool vs. standard static educational material on increasing HPV vaccination intent and uptake among female university students aged 18-26.

ELIGIBILITY:
Inclusion Criteria:

* enrolled at the University of Michigan

Exclusion Criteria:

* receipt of any doses of HPV vaccine

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 661 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Determine the effect of the MeFirst tool, a tailored, online HPV vaccination decision-making guide, on HPV vaccination intention and/or uptake. | Immediately post intervention, 3 months and 12 months
  Intention will be assessed on a five-point scale immediately after and at 3 and 12 months. Uptake will be assessed by yes/no/don't know response to the statement, "I have received at least 1 dose of the HPV vaccine" at 3 and 12 months.

SECONDARY OUTCOMES:
Determine the effect of the MeFirst tool on HPV-related knowledge. | Immediately post intervention, 3 months and 12 months
  Comparing 5 or 10-point scales measuring participants' HPV-related knowledge (HPV, HPV vaccination, and cervical cancer) immediately post-intervention and at 3 months and 12 months.

OTHER OUTCOMES:
Determine acceptability of the MeFirst tool to participants. | Immediately post intervention, 3 months and 12 months
  Participants answer five 5-point scale questions about the acceptability of the MeFirst tool immediately post intervention, and at 3 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa K Dalton, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Univeristy of Michigan, Ann Arbor, Michigan, United States